CLINICAL TRIAL: NCT06239233
Title: Gallbladder Infundibulum as a Guide for Ductal Identification in Laparoscopic Cholecystectomy in Nepalese Population at Tertiary Care Hospital
Brief Title: Gallbladder Infundibulum as a Guide for Ductal Identification.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nepal Mediciti Hospital (Other)
Responsible Party: Principal Investigator, Rajiv Mishra, Doctor, Nepal Mediciti Hospital
Other Study IDs: 427/2023
Record Dates: First submitted 2023-12-28; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Gallstone Disease
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — The surgeon makes small incisions in the abdominal wall, usually around the navel.
  Trocars (hollow tubes) are inserted through these incisions to provide access for the laparoscope and specialized instruments.
  A laparoscope, a thin tube with a light and camera, is inserted through one of the trocars. It allows the surgical team to visualize the abdominal cavity on a monitor.
  The surgeon carefully identifies the gallbladder and the cystic duct, which connects the gallbladder to the common bile duct.
  The cystic duct and artery are clipped and cut to disconnect the gallbladder from the biliary system. This step ensures the safe removal of the gallbladder.
  The surgeon gently detaches the gallbladder from the liver bed and removes it through one of the small incisions.
  Any bleeding vessels are sealed, and the small incisions are closed with stitches or surgical glue.

SUMMARY:
Introduction: Bile duct injury (BDI) is a catastrophic complication of cholecystectomy, and misidentification of the cystic anatomy is considered to be the main cause. Although several techniques have been developed to prevent BDI, such as the "critical view of safety", the infundibular technique, the rates remain higher during laparoscopic cholecystectomy (LC) than during open surgery. Strategy for ductal identification during laparoscopic cholecystectomy can help to prevent laparoscopic bile duct injury.

Methods: A prospective study of 196 patients who will undergo LC during the study period of one year at Nepal Mediciti Hospital will be conducted. The gallbladder infundibulum will be classified by its position located on an imaginary clock with the gallbladder neck as the center point of the dial, 3 o'clock position as cranial, 6 o'clock as dorsal, 9 o'clock as caudal, and 12 o'clock as ventral, as well as the axial position. Patient demographics, pathologic variables and infundibulum classification will be evaluated. Detailed analysis of ductal identification based on gallbladder infundibulum position will be performed in this study. All infundibulum positions will be recorded during intraoperative laparoscopic procedure.

DETAILED DESCRIPTION:
1. Objectives:

General Objective:

To investigate the potential association between infundibulum orientation and cystic duct identification during laparoscopic cholecystectomy.

Specific Objective:

1. To assess the influence of different infundibulum orientations on the success rate and time taken for cystic duct identification.
2. To evaluate the incidence and risk factors associated with post-operative morbidities following laparoscopic cholecystectomy.

Age, Sex, Ethnicity, Religion, Clinical Diagnosis, Intra operative gall bladder infundibulum orientation, relation of cystic duct with infundibulum, post operative complications. Success of cystic duct identification, duration of surgery, intraoperative blood loss and conversion to open are dependent variables and Position of infundibulum demographic, preoperative laboratory parameters, ultrasonographic findings are independent variables.

2. Ethical Considerations:

Ethical clearance was taken from National Health research council. Patient confidentiality and privacy will be maintained throughout the data collection and analysis process.

3. Data Collection:

Data will be collected on a structured Proforma covering the relevant subject matter of the study. A detailed orientation of the study and enrollment systems will be given to all doctor colleagues and ward in-charge for admitted patients. Upon receiving a case fulfilling the inclusion criteria, he/she will be given adequate explanation about the disease process, procedures performed and about the study. He/she will be assured of full confidentiality and would be asked if he/she wants to enroll in the study or not and an informed written consent taken subsequently. A detailed clinical history, clinical examination with appropriate investigations will be carried out. Demographic data will be collected including age, sex, and occupation. The relevant investigation including complete blood count, urine routine, blood sugar, blood urea, serum creatinine, serum electrolyte s, liver function test, chest X-ray including both dome of diaphragm, ECG ultrasonography of abdomen and pelvis etc. will be done as required for diagnosis. After establishing the diagnosis informed consent will be obtained. All patients diagnosed with gall stone disease will undergo laparoscopic cholecystectomy using three ports which will be performed under general anesthesia. First 10-millimeter port will be placed in infraumbilical region using open technique. Pneumoperitoneum will be created using carbon dioxide up to pressure of 12mm of Hg. Another 10-millimeter port will be placed in epigastrium below xiphoid process. Final 5-millimeter port will be placed in right hypochondrium. Adhesiolysis will be done if necessary. Visceral peritoneum over gall bladder infundibulum will be removed and Hartmann's pouch will be looked for.

Classification of the gallbladder infundibulum: The gallbladder infundibulum is variable in size and shape, and when this funnel-shaped portion is eccentrically inflated, it is called a Hartmann's pouch. According to our experience, this pouch lies at different directions with respect to the cystic duct and the common bile duct with a certain regularity. As the patient is placed in a supine position, and the surgeon stands on the left side of the patient with a line-of-sight from left to right, an imaginary clock facing the surgeon is vertically placed with the gallbladder neck as the center point of the dial. The Hartmann's pouch is assigned a location on this imaginary clock face to distinguish its positions (with the 3 o'clock position as cranial, 6 o'clock as dorsal, 9 o'clock as caudal, and 12 o'clock as ventral). In addition, if the infundibulum portion is uniformly dilated without a Hartmann's pouch, the investigators refer to this condition as axial position.

Furthermore, if the infundibulum with axial position is obviously inflated, it is defined as type I, otherwise, it is defined as type II(1). All the positions of the infundibulum will be identified during the laparoscopic process. Whether the Hartmann's pouch guide the investigator in finding the cystic duct will be noted. The time of surgery, blood loss, need for additional port placement and conversion to open will be noted.

4. Inclusion and Exclusion Criteria:

Inclusion criteria:

All the patient undergoing laparoscopic cholecystectomy for gall stone disease above age 18years.

Exclusion criteria:

Patients undergoing Laparoscopic cholecystectomy for Carcinoma Gallbladder. 5. Patient Consent:

Informed consent from patients for inclusion in the registry will be obtained, ensuring that they understand the purpose of the registry and the use of their data for research.

6. Data Quality and Validation:

Reliability of the study tool will be ensured by involving multiple observers and coming to an agreeable conclusion and as mentioned in methodology a complete standardized instructions about the tool will be employed. Validity of the study tool will be maintained by pilot testing and taking adequate sample to represent the population.

7. Statistical Analysis: Data management and analysis will be done in Excel and IBM SPSS 20. Tables, pie charts and bar diagrams will be used to demonstrate the results. Mean age (in years), Frequency and percentage of different sex, religion, occupation, co-morbidities, high total leukocyte count, abnormal renal function test, liver function test, will be calculated. Frequency and percentage of different position of infundibulum, success of cystic duct identification, conversion to open cholecystectomy will be calculated. Mean intraoperative blood loss (in milliliters), duration of operation time (in minutes), length of hospital stay (in hours) will be calculated. Frequency and percentage of post operative complications will be calculated. Logistic regression will be used to see any potential association between infundibulum orientation and success of cystic duct identification.

10. Dissemination: The results will be published in a peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* All the patient undergoing laparoscopic cholecystectomy for gall stone disease above age 18years.

Exclusion Criteria:

* Patients undergoing Laparoscopic cholecystectomy for Carcinoma Gallbladder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic cholecystectomy at Nepal Mediciti Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-10-19 (Estimated); Study Completion 2024-10-19 (Estimated)

PRIMARY OUTCOMES:
The investigator will identify the position of the Hartmann's pouch if present as 12,3,6 and 9 o' clock position. If the Hartmann's pouch is absent, then it will be labelled as axial type. Collected data will be aggregated in percentage. | 1 year.
  Primary outcome involves evaluating the effectiveness of the gallbladder infundibulum as a landmark for identifying and dissecting the bile ducts during the surgical procedure. The success rate could be measured by the proportion of cases in which the gallbladder infundibulum facilitated accurate and safe identification of the ductal structures.
  Number of participants with successful identification of cystic duct following Hartmann's pouch of Gall bladder infundibulum will be shown in percentage. Linear regression will be used to calculate the association between different position of infundibulum and sucess of identification of cystic duct.

SECONDARY OUTCOMES:
Incidence and risk factors associated with post-operative morbidities. | [Time Frame: 1 year]
  Incidence and risk factors for post-operative morbidities in laparoscopic cholecystectomy is crucial for improving patient outcomes, refining surgical techniques, and guiding preoperative counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Mishra, M.S., Principal Investigator — Nepal Mediciti Hospital
Locations (1):
- Nepal Mediciti Hospital, Kathmandu, Central, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shang P, Liu B, Li X, Miao J, Lv R, Guo W. A practical new strategy to prevent bile duct injury during laparoscopic cholecystectomy. A single-center experience with 5539 cases. Acta Cir Bras. 2020;35(6):e202000607. doi: 10.1590/s0102-865020200060000007. Epub 2020 Jul 8. PMID 32667588
- See also: A practical new strategy to prevent bile duct injury during laparoscopic cholecystectomy. A single-center experience with 5539 cases. — https://www.scielo.br/j/acb/a/TkX89kBjMPJQ74QDrBC558Q/?lang=en